CLINICAL TRIAL: NCT02379468
Title: Phase IIIb, A Prospective, Open Label, Randomized, Controlled, Parallel Group, Multicenter Clinical Trial of 3 Months Duration Comparing Topical Application of Royal Jelly and Panthenol (PEDYPHAR® Ointment) to Panthenol Ointment Only for Diabetic Foot Ulcers Treatment.
Brief Title: Efficacy & Safety of Pedyphar Ointment in Diabetic Foot Ulcer Treatment
Acronym: PEDFUT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Egyptian Pharmaceutical Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EEPI_ PED_001
Record Dates: First submitted 2015-02-19; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic; Foot; Ulcer
MeSH Terms: conditions — Diabetic Foot; Ulcer | interventions — dexpanthenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pedyphar (Experimental): Ointment
  Interventions: Drug: Pedyphar Ointment
- Panthenol (Active Comparator): Ointment
  Interventions: Drug: Panthenol

INTERVENTIONS:
Drug: Pedyphar Ointment
  Arms: Pedyphar
Drug: Panthenol — Ointment
  Arms: Panthenol

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Pedyphar® ointment in the healing of foot ulceration in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed and dated by study subject.
2. Male or Female patients.
3. Age is ≥18 years old and ≤ 70 years old.
4. Clinical diagnosis of Diabetes Mellitus Type I or II with diabetic foot ulcer. A past history of Diabetes Mellitus and/or the use of anti-diabetic medications for the treatment of Diabetes Mellitus with diabetic foot ulcer are sufficient.
5. Presence of 1 or more DFU, less than 15 cm in its biggest diameter, with a Texas University grade ≤ 2 and ≤ grade 2 according to the Wagner Grading system.
6. Diabetic foot ulcer has been present for at least 4 weeks and no more than 2 years prior to screening.
7. If there is Diabetic Foot Ulcer Infection, It must be:

   1. Mild ( Presence of ≥ 2 manifestations of inflammation (purulence, or erythema, pain, tenderness, warmth, or indurations),any cellulitis/erythema extending ≤ 2 cm around the ulcer, and infection is limited to the skin or superficial subcutaneous tissues; no other local complications or systemic illness).

      Or:
   2. Moderate Infection (as above) in a patient who is systemically well and metabolically stable but which has ≥1 of the following characteristics: cellulitis extending >2 cm, lymphangitic streaking, spread beneath the superficial fascia, deep-tissue abscess, gangrene, and involvement of muscle, tendon, joint or bone.
8. If subject is female and of childbearing potential, she agrees to use a medically acceptable physical barrier method contraceptive during the treatment phase.
9. Be willing and able to participate in the study as an outpatient, make the required visits to the study center during the treatment periods, and comply with study requirements.
10. Receiving medical care for diabetes.

Exclusion Criteria:

1. DFU with a Texas score >2 and > grade 2 according to the Wagner Grading system.
2. Severe Infected DFU with clinical or para-clinical findings suggesting osteomyelitis (Infection in a patient with systemic toxicity or metabolic instability (e.g., fever, chills, tachycardia, hypotension, confusion, vomiting, leukocytosis, acidosis, severe hyperglycemia, or azotemia)
3. Clinically defined and documented severe arterial disease.
4. History of radiation therapy to the ulcer site.
5. If the study subject has Foot Ulcer of no diabetic pathophysiology.
6. Receiving corticosteroids or immune suppressive agents.
7. History of immune-vascular disease.
8. Known hypersensitivity to any component of Pedyphar® or Panthenol.
9. Patients undergoing hemodialysis.
10. Insufficient blood supply to Lower Limb (ankle-brachial index < 0.9).
11. Clinical findings suggesting complicated venous insufficiency of LL. Edema [Hyper pigmentation, Venous dermatitis, Chronic cellulitis, Cutaneous infarction (atrophie blanche), Ulceration]
12. Received treatment with any other investigational drug or device within the last 30 days
13. Unable to comply with the procedures described in the protocol
14. History of moderate to severe ischemic heart disease or any history of congestive heart failure, or has had a myocardial infarction within the previous 6 months.
15. Patients with a history of major hematological, renal or hepatic abnormalities.
16. Mentally or neurologically disabled patients that are considered not fit to approve their participation in the study.
17. Refusal to give informed consent.
18. Pregnant or Breastfeeding subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Percentage of diabetic patients with successful healing of foot ulceration in treated with Pedyphar® ointment | 12 weeks
  Efficacy
Time to complete wound healing within 12 weeks before the end of treatment duration. | 12 weeks

SECONDARY OUTCOMES:
To evaluate the healing process of Diabetic foot ulcer using Pedyphar® ointment compared with Panthenol ointment regarding changes of foot ulcer dimensions from baseline visit to the end of the study. | 12 weeks
To identify the reasons of treatment failure and delayed response | 12 weeks
To identify adverse events associated with the application of Pedyphar® ointment. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Samir H. Asaad, Prof., Principal Investigator — Alexandria University
Locations (4):
- Egypt (4):
  - Alexandria University, Alexandria, Alexandria Governorate
  - Tanta University, Tanta, Please Select
  - Ain Shames University, Cairo
  - Suez Canal University, Suez